CLINICAL TRIAL: NCT04056507
Title: Retrospective Study of Splenic Immunological Markers as Predictive Factors for Response to Splenectomy in Adult Patients Affected by a Immune Thrombocytopenic Purpura
Brief Title: Immunological Markers in Adult Patients With Immune Thrombocytopenic Purpura
Acronym: SPLENOTIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHU BX 2011/05
Record Dates: First submitted 2019-08-13; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Immune Thrombocytopenic Purpura; Splenectomy; Status
Keywords: Immunological parameters; Histological parameters
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — This work is done on frozen female rats of already splenectomized adult ITP patients. A notice of no objection will be asked to patients for permission to work on this frozen material. Similarly, 10 control rats, from patients who had had a splenectomy at Bordeaux University Hospital following a road accident, will be analyzed and compared to those of the patients. It is a work of immuno-marking on splenic tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ITP group: On frozen spleens of already splenectomized adult ITP patients.
  Interventions: Procedure: Immunolabeling
- Control group: On frozen control spleens from patients who had a splenectomy at the Bordeaux University Hospital following a road accident.
  Interventions: Procedure: Immunolabeling

INTERVENTIONS:
Procedure: Immunolabeling — Immunolabeling of abnormalities observed by the cell study in flow cytometry.

SUMMARY:
The aim of this study is to determine histological immunological parameters, sought on splenectomy pieces that may explain the failure or success of splenectomy in patients with ITP who had a splenectomy to treat their ITP(Immune thrombocytopenic purpura).

DETAILED DESCRIPTION:
Immune thrombocytopenic purpura (ITP) is a rare autoimmune thrombocytopenia whose incidence is 2 to 5 cases / 100,000 inhabitants / year. The potentially serious haemorrhagic risk is the major issue of management. A recent international consensus conference classifies PTI according to the duration of thrombocytopenia: acute ITP (<3 months), persistent ITP (3-12 months) and chronic ITP (> 12 months) (Rodeghiero 2009). In the acute or persistent phase, polyvalent immunoglobulins (IVIG) and / or corticosteroids are proposed. In the chronic phase, splenectomy is a possible cure for 70% of patients. No predictor of treatment response is known.

The pathophysiology of ITP is multifactorial: platelet phagocytosis, mediated by autoantibody, macrophages of the reticuloendothelial system, and destruction in the spleen, genetic background and / or environmental factor favoring the role of certain lymphocyte subpopulations, cytotoxic or regulatory T, via their cytokine environment, abnormalities of thrombopoiesis.

At present, no predictive factor of splenectomy success has been identified. The aim of this study is to determine histological immunological parameters, sought on splenectomy pieces that may explain the failure or success of splenectomy in patients with ITP who had a splenectomy to treat their ITP.

ELIGIBILITY:
Inclusion Criteria:

* The analyzed spleens belong to the collection of biological samples declared to the ministry by the Laboratory of Pathology of Haut-Lévêque Hospital (Dr Parrens).

Exclusion Criteria:

* Opposition of the patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Spleens come from patients with ITP (defined as thrombocytopenia <100 G / L) after an infectious, drug, autoimmune disease, hematological malignancy or immunodeficiency cause has been eliminated. Rodeghiero, 2009) who received a splenectomy to treat their condition in the department of Professor JL Pellegrin.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-04-12 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR) after splenectomy. | At the inclusion
  Determination of ITP status following Rodeghiero criteria : complete remission if platelet count > 100 G/L. patient who is not on complete remission after splenectomy will be considered to be failing.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François VIALLARD, Pr, Principal Investigator — University Hospital, Bordeaux